CLINICAL TRIAL: NCT06024122
Title: Brain Development in Young Children Following Mild Traumatic Brain Injury - Pilot Study
Acronym: KAOUENN
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Institut National de Recherche en Informatique et en Automatique (Other)
Responsible Party: Sponsor
Other Study IDs: C22-48; 2022-A02619-34 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-07-07; First posted 2023-09-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: TBI (Traumatic Brain Injury)
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with a mTBI: Children with a mTBI aged 3 to 5 years (i.e., up to 71 months and 31 days, i.e., before the 6th birthday) recruited from the paediatric emergency department of Rennes University Hospital.
  Interventions: Other: IRM exam
- Control with an orthopaedic injury: Children with an orthopaedic injury aged 3 to 5 years (i.e., up to 71 months and 31 days, i.e., before the 6th birthday) recruited from the paediatric emergency department of Rennes University Hospital.
  Interventions: Other: IRM exam

INTERVENTIONS:
Other: IRM exam — A non-sedated MRI scan will be performed to assess the structure and function of the children's brains

SUMMARY:
Concussions (also known as mild traumatic brain injury) are common in young children. In some children, they can lead to short- and long-term difficulties. However, our knowledge of the exact consequences of injuries on young children's brains and behavior is limited. These consequences may be different in children under 6, as their brains are fragile and undergoing significant developmental changes.

The aim of this study is to determine the extent to which a concussion sustained before the age of 6 years is associated with changes in young children's brain structure, function and behaviours, using a brain imaging.

In this study, the results of a group of 30 children with a concussion will be compared to those of 30 children of the same age with an orthopaedic injury to the upper or lower limbs.

ELIGIBILITY:
Inclusion Criteria:

* Patient group with mild traumatic brain injury (mTBI) :

  1. Children aged between 36 months (3 years) and 71 months and 31 days (5 years; before their 6th birthday)
  2. Presentation to the emergency department within 48 hours post-injury
  3. Documented, unintentional traumatic event (e.g. blow, fall, etc.) resulting in non-penetrating head injury
  4. Diagnosis of mTBI (World Health Organization (WHO) paediatric diagnostic criteria)
* Control group with orthopaedic injury:

  1. Children aged between 36 months (3 years) and 71 months and 31 days (5 years; before their 6th birthday)
  2. Presentation to the emergency department within 48 hours post-injury
  3. Documented, unintentional traumatic event (e.g. blow, fall, etc.) resulting in trauma to an upper or lower limb
  4. Diagnosis of simple fracture, sprain, contusion or unspecified trauma to a limb (mild).

Exclusion Criteria:

* Diagnosis of previous TBI (any severity, any age)
* Intentional injury,
* Administration of sedative drugs that can alter brain function
* Complications following injury
* MRI contraindication,
* Parent non-fluent in French,
* Prematurity,
* Diagnosis of a severe neurological, developmental, or psychiatric disorder
* Children in foster care at the time of recruitment

Ages: 36 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged between 36 months (3 years) and 71 months and 31 days (5 years; before their 6th birthday) with mTBI.
  Children aged between 36 months (3 years) and 71 months and 31 days (5 years; before their 6th birthday) with orthopaedic injury (simple fracture, sprain, contusion or unspecified trauma to a limb (mild))
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Persistent brain structure alterations | 3 months post-injury
  Quantitative assessment of the brain morphometry extracted from T1-w MRI sequence

SECONDARY OUTCOMES:
Persistent brain lesions - Volume | 3 months post-injury
  Volume of brain lesions measured with susceptibility MRI
Persistent brain lesions - Number | 3 months post-injury
  Number brain lesions measured with susceptibility MRI
Cerebral blood flow alteration | 3 months post-injury
  Cerebral blood flow quantified by arterial spin labelling perfusion MRI (ASL)
Functional integrity of brain networks | 3 months post-injury
  Functional connectivity (i.e., correlation between the activation of brain regions) measured by resting-state functional MRI
Structural integrity of brain networks | 3 months post-injury
  White matter micro-structure measured by diffusion MRI

OTHER OUTCOMES:
Acute and persistent post-concussive symptoms | Through study completion, an average of 3 months
  Assessment of post-concussive symptoms using the REACTIONS questionnaire
Persistent behavioural difficulties | 3 months post-injury
  Assessment of behaviour using the Strengths and Difficulties Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Fanny DÉGEILH, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Unité des urgences médicochirurgicales CHU Rennes, Rennes, France